CLINICAL TRIAL: NCT05070624
Title: Connecting Caregivers: A Randomized Controlled Trial to Evaluate Virtual Peer-Support for Family Caregivers of Individuals With Neuromuscular Disease
Brief Title: The Peer Support Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Reshma Amin, Associate Professor, The Hospital for Sick Children
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: CTO-3590
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Neuromuscular Diseases
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): After informed consent, we will assign participants in a 1:1 ratio to the intervention or control group using Randomize.net.
  Participants randomized to intervention group will get access to the Virtual Peer Support Program.
  Interventions: Behavioral: The Virtual Peer Support Program
- Control (No Intervention): Control group: Those randomized to the waitlist control will be given access to the peer support intervention on completion of the first 12-week program. A waitlist control group is an ethical alternative to no-treatment control groups when studying psychological and behavioral interventions 21. will have access to informational resources via the aTouchAway™ App and will also receive the intervention at the end of the trial.

INTERVENTIONS:
Behavioral: The Virtual Peer Support Program — Training: We have previously developed and beta-tested a virtual peer mentor training program adapted from the St. Jude's Research Hospital's (Memphis, USA) program for FCs of children with cancer for adults using HMV. Content & Design of the Virtual Peer-Support Program: The program will be delivered by the aTouchAway™ App used for the LIVE program. Participants will be requested to access peer mentors ≥1 time/week. Participants can choose to interact with a peer mentor which will be assigned as well as other peer participants. Onboarding: Participants and mentors will create a personal profile of their caregiving situation (e.g., duration of care, family member age and diagnosis), to enable selection of mentors by the research team believed to be well suited to address support needs, questions, and concerns based on similar lived experience.
  Arms: Intervention

SUMMARY:
Competent family caregivers (FC) are essential for successful caring for individuals with NMD. However, family caregiving is known to contribute to significant FC burden and social isolation, and negatively affects FC health. Infrastructure to support FCs is paramount to ensure that individuals with NMD can safely remain at home. Individuals with NMD have complex health problems, require a lot of care and they use the healthcare system often. COVID-19 physical distancing has increased the care burden and social isolation for many FCs. Infrastructure to support FCs is paramount to ensure that individuals with NMD can safely remain at home. Peer support includes emotional and informational support by an individual that has experienced a similar health problem. It improves health-related quality of life, increases self-efficacy and empowerment, and decreases stress in various patient and caregiver populations. With our study we plan to educate and empower individuals with NMD and their caregivers and develop a comprehensive peer support program.

ELIGIBILITY:
Eligibility Criteria for Peer-Support Program:

Inclusion Criteria

1. FC of individual with NMD that lives in Canada;
2. Speaks and reads English;
3. Access to internet and computer/tablet.

Exclusion Criteria:

We will exclude those Ventilator Assisted Individuals (VAI) and caregivers, who are:

1. Unable to communicate verbally in English
2. No access to internet and computer/tablet.

Eligibility Criteria for Peer Mentors:

Inclusion Criteria:

1. Criteria 1-3 above;
2. Completion of virtual peer support training;
3. Identified by the HMV team or self-referral.

Exclusion Criteria:

We will exclude those VAIs and caregivers, who are:

1. Unable to communicate verbally in English
2. No access to internet and computer/tablet.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Family Caregiver (FC) mastery measured using the Pearlin Mastery Scale (PMS) | baseline
  FC mastery measured using the Pearlin Mastery Scale (PMS) (Pearlin Mastery Scale;(scores range up to 28, higher scores = higher mastery) at baseline,
Family Caregiver (FC) mastery measured using the Pearlin Mastery Scale (PMS) at12 weeks | 12 week
  (FC) mastery measured using the Pearlin Mastery Scale (PMS) at12 weeks (Pearlin Mastery Scale; (scores range up to 28, higher scores = higher mastery)
Family Caregiver (FC) mastery measured using the Pearlin Mastery Scale (PMS) at 24 weeks | 24 week
  (FC) mastery measured using the Pearlin Mastery Scale (PMS) at 24 weeks (Pearlin Mastery Scale; (scores range up to 28, higher scores = higher mastery)

SECONDARY OUTCOMES:
Caregiver Competency - measured using the Caregiving Competence Scale | Baseline
  Caregiver Competency - measured using the Caregiving Competence Scale, The total scores of this 4-item scale ranged from 4 to 16, with higher scores indicating higher levels of caregiving competence
Caregiver Competency - measured using the Caregiving Competence Scale | 12 week
  Caregiver Competency - measured using the Caregiving Competence Scale, The total scores of this 4-item scale ranged from 4 to 16, with higher scores indicating higher levels of caregiving competence
Caregiver Competency - measured using the Caregiving Competence Scale | 24 week
  Caregiver Competency - measured using the Caregiving Competence Scale, The total scores of this 4-item scale ranged from 4 to 16, with higher scores indicating higher levels of caregiving competence
Family Caregiver Burden and Stress - measured using the Zarit Burden Interview | Baseline
  Family Caregiver Burden and Stress - measured using the Zarit Burden Interview (scores range up to 88, higher scores = higher burden)
Family Caregiver Burden and Stress - measured using the Zarit Burden Interview | 12 week
  Family Caregiver Burden and Stress - measured using the Zarit Burden Interview scores range up to 88, higher scores = higher burden)
Family Caregiver Burden and Stress - measured using the Zarit Burden Interview | 24 week
  Family Caregiver Burden and Stress - measured using the Zarit Burden Interview scores range up to 88, higher scores = higher burden)
Family Caregiver Depression and Anxiety: measured using the Depression and Anxiety Stress Scale | Baseline
  Family Caregiver Depression and Anxiety: measured using the Depression and Anxiety scores range up to 42, higher scores = higher depression and Anxiety)Stress Scale
Family Caregiver Depression and Anxiety: measured using the Depression and Anxiety Stress Scale | 12 week
  Family Caregiver Depression and Anxiety: measured using the Depression and Anxiety scores range up to 42, higher scores = higher depression and Anxiety)Stress Scale
Family Caregiver Depression and Anxiety: measured using the Depression and Anxiety Stress Scale | 24 week
  Family Caregiver Depression and Anxiety: measured using the Depression and Anxiety scores range up to 42, higher scores = higher depression and Anxiety)Stress Scale
Family Caregiver Experience of the virtual peer support explored using qualitative interviews. | Baseline
  Family Caregiver Experience of the virtual peer support explored using qualitative interviews.
Family Caregiver Experience of the virtual peer support explored using qualitative interviews. | 12 week
  Family Caregiver Experience of the virtual peer support explored using qualitative interviews.
Family Caregiver Experience of the virtual peer support explored using qualitative interviews. | 24 week
  Family Caregiver Experience of the virtual peer support explored using qualitative interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Reshma Amin, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No